CLINICAL TRIAL: NCT03520348
Title: Phase I Clinical Study, to Evaluate the Safety and Tolerability of the Ophthalmic Gel PRO-167 Versus Corneregel®, on the Ocular Surface of Ophthalmological and Clinically Healthy Subjects.
Brief Title: Safety and Tolerability of the Ophthalmic Gel PRO-167 Versus Corneregel® on Healthy Subjects.
Acronym: PRO-167/I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOPH167-0816/I
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye; Dry Eye Syndrome of Unspecified Lacrimal Gland
Keywords: dry eye; eye lubricants; eye lubricant gel; PRO-167
MeSH Terms: conditions — Dry Eye Syndromes | interventions — dexpanthenol

STUDY DESIGN:
Intervention Model Description: Phase I clinical trial, controlled, of parallel groups, double blind, randomized, exploratory.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The blinding will correspond to the research subject and the principal investigator. In addition, the statistical analysis will be carried out in a blinded manner for the partial and final analysis.
  The masking will be done using boxes in the primary packaging identical in the two groups. Blinding for the research subject and the researcher will be done by replacing the commercial labels in the case of the comparator in the bottles and the use of identical labels that contain the allocation number.
  Blinding may be opened in the following cases:
  1. Presence of a serious adverse event.
  2. Safety alarm due to the use of the drugs under study.
  3. In case the sponsor determines it for any reason of security or other reason that considers pertinent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-167 (Experimental): Dose: a strip approximately 1 cm long, 4 times a day during the period of vigil, in the bottom
  Interventions: Drug: PRO-167
- Corneregel® (Active Comparator): Dose: a strip approximately 1 cm long, 4 times a day during the period of vigil, in the bottom of the right eye sac.
  Interventions: Drug: Corneregel

INTERVENTIONS:
Drug: PRO-167 — Dexpanthenol 5%. Ophthalmic gel produced by Laboratorios Sophia, S.A. of C.V., Zapopan, Jalisco, Mexico.
  Route of administration: ophthalmic
  Other Names: dexpanthenol
  Arms: PRO-167
Drug: Corneregel — Dexpanthenol 5%. Ophthalmic gel developed by Bausch and Lomb, Berlin, Germany. Route of administration: ophthalmic
  Other Names: dexpanthenol
  Arms: Corneregel®

SUMMARY:
Title of the study:

Phase I clinical trial, to evaluate the safety and tolerability of the ophthalmic gel PRO-167 versus Corneregel®, on the ocular surface of ophthalmological and clinically healthy subjects.

Methodology:

Phase I clinical trial, controlled, of parallel groups, double blind, randomized, exploratory.

Goals:

To evaluate the safety and tolerability of the ophthalmic gel PRO-167 manufactured by Laboratorios Sophia S.A. of C.V. on the ocular surface of clinically healthy subjects.

Hypothesis:

Ophthalmic gel PRO-167 has a safety and tolerability profile similar to that of its comparator in healthy subjects.

DETAILED DESCRIPTION:
Therapeutic indication:

Corneal surface reepithelizing

Statistical methodology:

The data will be expressed with measures of central tendency: mean and standard deviation for the quantitative variables. The qualitative variables will be presented in frequencies and percentages. The statistical analysis will be carried out through the Mann-Whitney U test for quantitative variables. The difference between the qualitative variables will be analyzed by means of square chi (Chi2). An alpha ≤ 0.05 will be considered significant.

Study period:

3 to 4 months

Development phase: I

Number of patients:

24 subjects, divided into 2 groups (12 eyes exposed per group)

Test product, dose and route of administration, lot number:

PRO-167. Dexpanthenol 5%. Ophthalmic gel produced by Laboratorios Sophia, S.A. de C.V., Zapopan, Jalisco, Mexico.

* Dose: a strip approximately 1 cm long, 4 times a day during the period of vigil, in the bottom of the right eye sac.
* Route of administration: ophthalmic.

Reference product, dose and route of administration, lot:

* Corneregel. Dexpanthenol 5%. Ophthalmic gel developed by Bausch and Lomb, Berlin, Germany.
* Dose: a strip approximately 1 cm long, 4 times a day during the period of vigil, in the bottom of the right eye sac.
* Route of administration: ophthalmic

Evaluation criteria:

Primary security outcome variable:

- Density of goblet cells.

Secondary security variables:

* Epithelial defects in cornea and conjunctiva.
* Presence of adverse events.

Secondary outcome variables:

* Intraocular pressure.
* Visual ability
* Break time of the tear film.

Outcome variables of tolerability:

* Burning.
* Foreign body sensation.
* Itching.
* Eye comfort index.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Systemically and ophthalmologically healthy subjects evaluated during the clinical history.
* Age between 18 to 45 years.
* Both genders.
* Blood tests [complete blood count, blood chemistry of three elements and liver function tests within normal parameters specified by the reference laboratory with a lower and upper margin of 10%.
* Vital signs within normal parameters.
* Visual capacity 20/30 or better, in both eyes.
* Intraocular pressure ≥11 and ≤ 21 mmHg.

Exclusion Criteria:

* Subjects with a history of hypersensitivity to any of the components of the research products.
* Subject users of topical ophthalmic medications of any pharmacological group.
* Subject users of medication by any other route of administration.
* Women who are pregnant or breastfeeding.
* Women without a history of hysterectomy, oophorectomy, who do not ensure a hormonal contraceptive method or intrauterine device during the study period.
* Subjects with participation in clinical research studies 90 days prior to inclusion in the present study.
* Diagnosis of liver disease or triple the normal upper value of any of the following liver enzymes: aspartate transferase (AST), alanine transferase (ALT) or bilirubin.
* Inability to attend or answer the evaluations made in each of the visits.
* Positive smoking (specified as cigarette consumption regardless of quantity and frequency)
* Positive alcoholism (specified as the consumption of alcoholic beverages, regardless of quantity and frequency, during the study intervention period)
* Contact lens users

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Centro Oftalmológico San Angel, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Villegas P, Navarro-Sanchez AA, Sanchez-Rios A, Olvera-Montano O, Baiza-Duran LM. Reexamining Ophthalmic Drugs, Safety and Tolerability in Phase 1 Clinical Trials. Ther Clin Risk Manag. 2021 Oct 21;17:1123-1134. doi: 10.2147/TCRM.S331294. eCollection 2021. PMID 34707360

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-167: Dose: a strip approximately 1 cm long, 4 times a day during the period of vigil, in the bottom
  PRO-167: Dexpanthenol 5%. Ophthalmic gel produced by Laboratorios Sophia, S.A. of C.V., Zapopan, Jalisco, Mexico.
  Route of administration: ophthalmic
- Corneregel®: Dose: a strip approximately 1 cm long, 4 times a day during the period of vigil, in the bottom of the right eye sac.
  Corneregel: Dexpanthenol 5%. Ophthalmic gel developed by Bausch and Lomb, Berlin, Germany.
  Route of administration: ophthalmic
Period: Overall Study
Arm/Group | PRO-167 | Corneregel®
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: clinically and ophthalmologically healthy subjects
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-167 | Corneregel® | Total
Number analyzed (Participants) | 12 | 12 | 24
Number analyzed (eyes) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.25 (6.84) | 28.17 (4.95) | 28.71 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Goblet Cell Density (GCD)
Description: the cells will be measured per square millimeter, it is a continuous variable taken by means of cytology per impression, the normal value is higher than 500 cells per square millimeter
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
cells/mm^2 | 444 (112.5) | 440 (127.2)
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — It is considered less than 20% of differences between groups to consider non-inferiority; p = 0.285, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Presence of Adverse Events (EAS)
Description: the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent.
Time Frame: during the 11 days of evaluation, including the safety call (day 13).
Measure: Number; unit: cases
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
cases | 7 | 6
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — it is considered noninferiority if there are no differences in the 20% between the research drug and the reference medicine; p = 0.680, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Intraocular Pressure (IOP)
Description: the intraocular pressure will be evaluated by means of the Goldman applanation tonometry whose unit of measurement is millimeters of mercury (mmHg), it is a continuous variable and its normality range is between 11 - 21 mmHg
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
mmHg | 13.14 (2.22) | 13.56 (1.99)
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.839, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Breakup Time (BUT)
Description: breakup time lacrimal film is a continuous variable that will be measured in seconds, evaluating the time it takes to break it, is done by direct counting and the normality range greater than 10 seconds.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
seconds | 8.92 (2.1) | 7.75 (2.1)
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.137, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Chemosis
Description: The chemosis will be evaluated, as a nominal variable, by direct observation and it will be staged as present and absent, where the normality is that said variable is absent.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
cases | 0 | 0

6. Secondary Outcome: Ocular Burning (OB)
Description: ocular burning is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale: Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.Frequency: At all times, almost at all times, 50% of the time, almost in no time, at any time. where the normality of the frequency is in no time.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
percentage of participants
  Absent | 66.7 | 75
  mild | 29.2 | 16
  moderate | 4.2 | 8.3
  Severe | 0 | 0
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.667, Chi-squared, Corrected

7. Secondary Outcome: Epithelial Defects (ED)
Description: The epithelial defects will be evaluated by means of two stains, green lissamine, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the oxford scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
cases
  grade 0 | 8 | 8
  grade I | 4 | 3
  grade II | 0 | 1
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.561, Chi-squared, Corrected

8. Secondary Outcome: Conjunctival Hyperemia (CH)
Description: Conjunctival hyperemia will be evaluated as an ordinal variable, by direct observation and staged using the Efron scale as Normal / Very Light / Mild / Moderate / Severe. Based on this scale, the normal and mild stages are considered without pathologies or normal. Mild, moderate and severe are considered pathological.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
percentage of participants
  Normal | 16.7 | 8.3
  Very mild | 66.6 | 66.7
  Mild | 16.7 | 25
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 1.000, Chi-squared

9. Secondary Outcome: Foreign Body Sensation (FBS)
Description: Foreign body sensation is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.
  Frequency: At all times, almost at all times, 50% of the time, almost in no time, at any time. where the normality of the frequency is in no time.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
percentage of participants
  Absent | 79.2 | 91.7
  Very mild | 20.8 | 8.3
  Mild | 0 | 0
  Moderate | 0 | 0
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.317, Chi-squared, Corrected

10. Secondary Outcome: Ocular Pruritus (P)
Description: Ocular pruritus is a nominal variable that will be evaluated by direct questioning to the research subject, then it will be staged according to the following scale:
  Severity: Absent, very mild, mild, moderate and severe, where the normality of severity is absent.
  Frequency: At all times, almost at all times, 50% of the time, almost in no time, at any time. where the normality of the frequency is in no time.
Time Frame: will be evaluated at the end of the treatment at the final visit (day 11)
Population: the statistical analysis of the sample was carried out by protocol
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | PRO-167 | Corneregel®
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 24 | 24
percentage of participants
  Absent | 41.7 | 66.7
  Very mild | 50 | 16.7
  Mild | 8.3 | 16.7
  Moderate | 0 | 0
Statistical Analysis 1: Comparison: PRO-167 vs Corneregel®; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.414, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for a total of 13 days, including the scrutiny visit (day 0) until the safety call (day 13)
Arm/Group | PRO-167 | Corneregel®
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-167 (N=12) | Corneregel® (N=12)
headache (General disorders) | 2 (2) | 1 (1)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
earache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
dysgeusia (Gastrointestinal disorders) | 0 (0) | 1 (1)
non-infectious diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1)
eyelid bruise (Eye disorders) | 1 (1) | 0 (0)
Ocular burning (Eye disorders) | 4 (4) | 3 (3)
elevated liver enzymes (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Researchers can not disseminate research results unless they obtain written authorization from the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03520348/Prot_SAP_000.pdf